CLINICAL TRIAL: NCT00254813
Title: Fast Titration Of Quetiapine Versus Currently Approved Titration: A Randomised, Multicentre, Parallel Group Open Trial In Schizophrenia And Schizoaffective Disorder
Brief Title: Fast Titration Of Quetiapine Versus Currently Approved Titration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1449L00003
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Psychotic Disorders
Keywords: Schizophrenia; Schizoaffective disorder
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a more rapid dose titration in acute schizophrenic patients compared to the conventional titration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, male or female between 18 and 60 years old, having acute exacerbation of their schizophrenia or schizoaffective disorder requiring admission to hospital. Should stay in hospital for at least 7 days.

Exclusion Criteria:

* Patients treated with Risperdal consta or Clozapine last 28 days, pregnancy or breast-feeding, patients known to be intolerant or unresponsive to quetiapine, known arrhythmia, other serious medical conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2004-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with moderate and severe adverse events

SECONDARY OUTCOMES:
Mean daily level of somnolence and orthostatic dizziness as rated on AE intensity scale

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Norway Medical Director, MD, Study Director — AstraZeneca
Locations (7):
- Norway (7):
  - Research Site, Arendal
  - Research Site, Ålesund
  - Research Site, Klepp stasjon
  - Research Site, Kristiansand
  - Research Site, Nesttun
  - Research Site, Oslo
  - Research Site, Ottestad